CLINICAL TRIAL: NCT05824988
Title: Drug Exposure and Minimum Inhibitory Concentration in the Treatment of Mycobacterium Avium Complex Lung Disease: a Prospective Observational Cohort Study
Brief Title: Drug Exposure and Minimum Inhibitory Concentration in the Treatment of MAC Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Fudan University (Other); University of Sydney (Other); Karolinska Institutet (Other); Shanghai Municipal Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Wei Sha MD & PhD, Director of Clinic and Research Center of Tuberculosis, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: K22-149Z
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Mycobacterium Avium Complex; Mycobacterium Avium-Intracellulare Infection; Gram-Positive Bacterial Infections; Mycobacterium Infections
Keywords: Treatment; Minimum Inhibitory Concentration; Drug Concentration; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; Gram-Positive Bacterial Infections; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mycobacterium avium complex isolates will be frozen and stored for whole genome sequencing in order to explore development of drug resistance-conferring mutations and to distinguish relapse from reinfection. Blood samples will be collected and stored for drug concentration analysis.

GROUPS / COHORTS (1):
- Patients with MAC lung disease
  Interventions: Other: Drug exposure

INTERVENTIONS:
Other: Drug exposure — Drug concentrations will be measured after one-month antimycobacterial treatment. Area under drug concentration-time curve (AUC) and maximum concentration (Cmax) will be calculated.

SUMMARY:
The incidence and prevalence of nontuberculous mycobacteria (NTM) infections have gradually increased over the years worldwide (1-3). In China, Mycobacterium avium complex (MAC) was the most prevalent NTM specie (4), while challenged by long treatment duration, frequent drug-induced adverse events, lack of treatment alternatives, poor treatment outcome and high recurrence rate (5, 6). In order to maximize the efficacy of the few available drugs and prevent the development of drug resistance, ensuring adequate plasma drug concentrations are of importance. Despite the role of pathogen susceptibility, determined by minimum inhibitory concentration (MIC), is non-negligible, the evidences regarding its association with treatment outcome are limited, especially for rifamycin and ethambutol. The difficulties in explaining the clinical values of MIC might partially be attributed to the lack of in vivo drug exposure data, which cannot be accurately predicted by the dose administered because of between-patient pharmacokinetic variability (7). Therapeutic drug monitoring (TDM) is a strategy to guide and personalize treatment by measuring plasma drug concentrations and pathogen susceptibility, which might have the potential to improve treatment response to MAC lung disease.

In this observational study, the hypothesis is that the drug exposure and/or MIC of antimycobacterial drugs are correlated to the treatment response of MAC lung disease, which is assessed from the perspective of treatment outcome, mycobacterial culture negative conversion, lung function, radiological presentation and self-reported quality of life. Consenting adult patients with culture-positive MAC lung disease will be recruited in study hospital. Respiratory samples (sputum and/or bronchoalveolar lavage fluid) will be collected regularly for mycobacterial culture on the basis of BACTEC MGIT 960 system and MIC will be determined using a commercial broth microdilution plate. Drug concentrations will be measured at 1 and/or 6 months after treatment initiation using liquid chromatography tandem mass spectrometry (LC-MS/MS). The final treatment outcome is recorded at the end of MAC treatment and defined according to an NTM-NET consensus statement (8).

DETAILED DESCRIPTION:
This is an observational cohort study conducted to enrol consenting adult patients with culture-positive MAC lung disease in study hospital (n=100). The diagnosis and treatment of MAC lung disease will adhere to the ATS/ERS/ESCMID/IDSA and Chinese national guidelines (9, 10). Patients treated with a regimen composed of macrolides, rifamycin and ethambutol at minimum are screened for eligibility. Detailed demographic, behaviour, clinical and laboratory information will be recorded at baseline. Respiratory samples (sputum and/or bronchoalveolar lavage fluid) will be collected at baseline and once every 3 months until treatment completion for mycobacterial culture using BACTEC MGIT 960. Time to mycobacterial culture positivity (TTP) will be recorded to estimate the bacterial load as an alternative for colony forming units count. MIC determination will be performed for baseline, six-month and/or the last available positive culture during treatment with the Sensititre™ SLOMYCO2 Susceptibility Testing Plate, to assess the development of acquired drug resistance.

Drug concentrations will be measured for all study patients at one month after treatment initiation. Rich blood sampling (0, 1, 2, 4, 6 and 8 hours after drug intake) will be implemented for the first 30 patients aged < 65 years to enable the development of population pharmacokinetic models. A limited sampling strategy (2 and 6 hours after drug intake) will be applied for the rest patients to increase the feasibility of study. Additional blood sampling will be given for patients with poor treatment response at six months with limited sampling strategy. The developed pharmacokinetic models will be used to accurately calculate the area under the plasma concentration versus time curve (AUC) and peak plasma concentration (Cmax), as the main exposure variables. To comprehensively assess the response to MAC treatment, mycobacterial culture, lung function test, computerized tomography (CT) scan and questionnaires for well-being will be taken regularly in this study. The final treatment outcome is recorded at the end of MAC treatment and defined according to an NTM-NET consensus statement (8). Post-treatment visits are given at 6 and 12 months after treatment completion to assess the recurrence of MAC lung disease.

Together with bacteria MIC and clinical data, the Cmax/MIC and AUC/MIC for antimycobacterial drugs will be explored to deepen our understandings on the correlation of pharmacokinetic and/or pharmacodynamic indices with treatment response, which may guide development of new dosing strategies.

ELIGIBILITY:
Inclusion Criteria:

* Culture-positive MAC lung disease
* MAC treatment at the Shanghai Pulmonary Hospital
* A regimen composed of at least the core drugs, i.e., macrolides, rifamycin and ethambutol, in doses not lower than recommended according to the ATS/ERS/ESCMID/IDSA and Chinese national guidelines
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Confirmed mixed infection with mycobacterial species, including M.tuberculosis and other NTM species
* Ongoing with any antimycobacterial treatment for more than one month, including tuberculosis and NTM
* Patients admitted to the intensive care unit
* Off-label use for any study drugs, such as inhalation of amikacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with and treated for MAC lung disease in study hospital in Shanghai, China will be screened for eligibility. Patients will be informed and asked to participate in the study both orally and in writing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) for key antimycobacterial drugs, separate and in relation to minimum inhibitory concentration | one-month of treatment
  Descriptive data of the distribution of Cmax for key antimycobacterial drugs in patients with MAC lung disease, with regard to existing recommended levels. Their associations with treatment response will be investigated.
Area under the plasma concentration versus time curve (AUC) for key antimycobacterial drugs, separate and in relation to minimum inhibitory concentration | one-month of treatment
  Descriptive data of the distribution of AUC for key antimycobacterial drugs in patients with MAC lung disease, with regard to existing recommended levels. Their associations with treatment response will be investigated.

SECONDARY OUTCOMES:
Proportion of patients with cure of MAC lung disease | 12-18 months
  The proportion of patients with cure of MAC lung disease at the end of treatment. The definition of treatment outcome will refer to an NTM-NET consensus statement, on the basis of mycobacterial culture as well as patient-reported and/or objective improvement of symptoms.
Six-month culture conversion | 6 months
  The proportion of patients with culture negative conversion after 6 months of MAC treatment.
Time to culture conversion | 12-18 months
  Time (in months) from start of treatment until the first out of three consecutive negative cultures, collected at least 30 days apart.
Proportion of patients with significant changes in drug resistance profile | 12-18 months
  The proportion of patients with significant changes in the drug resistance profile, phenotypic (MIC) and genotypic (whole genome sequencing) of the antimycobacterial drugs used, during MAC treatment.
Resolution of pulmonary lesions or cavitation | 12-18 months
  Resolution or deterioration of pulmonary lesions or cavitation during MAC treatment by CT scan.
Proportion of patients with improved forced expiratory volume in 1 second (FEV1) | 12-18 months
  Decrease or increase of FEV1 during MAC treatment by lung function test.
Proportion of patients with improved forced vital capacity (FVC) | 12-18 months
  Decrease or increase of FVC during MAC treatment by lung function test.
Proportion of patients with improved quality of life | 12-18 months
  Improvement or deterioration of quality of life during MAC treatment by the St. George's Respiratory Questionnaire (SGRQ). The SGRQ score ranges from 0 to 100, with higher scores indicating more limitations.
Proportion of patients with grade 3 or 4 adverse events | 12-18 months
  The proportion of patients with grade 3 or 4 adverse events during MAC treatment, according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) guidelines.
Number of patients with recurrence of MAC lung disease | 24-30 months
  The number of patients with recurrence of MAC lung disease within one year post treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Sha, MD, Prof, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Xubin Zheng, MPH, PhD, Study Director — Shanghai Pulmonary Hospital, Shanghai, China; Biao Xu, Prof, Study Chair — Fudan University; Jan-Willem Alffenaar, PhamD, Prof, Study Chair — University of Sydney; Judith Bruchfeld, Ass. Prof, Study Chair — Karolinska Institutet; Yi Hu, Ass. Prof, Study Chair — Fudan University; Lina Davies Forsman, MD, PhD, Study Chair — Karolinska Institutet; Yangyi Zhang, MPH, Study Chair — Shanghai Municipal Center for Disease Control and Prevention
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winthrop KL, Marras TK, Adjemian J, Zhang H, Wang P, Zhang Q. Incidence and Prevalence of Nontuberculous Mycobacterial Lung Disease in a Large U.S. Managed Care Health Plan, 2008-2015. Ann Am Thorac Soc. 2020 Feb;17(2):178-185. doi: 10.1513/AnnalsATS.201804-236OC. PMID 31830805
- [Background] Lee H, Myung W, Koh WJ, Moon SM, Jhun BW. Epidemiology of Nontuberculous Mycobacterial Infection, South Korea, 2007-2016. Emerg Infect Dis. 2019 Mar;25(3):569-572. doi: 10.3201/eid2503.181597. PMID 30789139
- [Background] Ringshausen FC, Wagner D, de Roux A, Diel R, Hohmann D, Hickstein L, Welte T, Rademacher J. Prevalence of Nontuberculous Mycobacterial Pulmonary Disease, Germany, 2009-2014. Emerg Infect Dis. 2016 Jun;22(6):1102-5. doi: 10.3201/eid2206.151642. PMID 27191473
- [Background] Tan Y, Deng Y, Yan X, Liu F, Tan Y, Wang Q, Bao X, Pan J, Luo X, Yu Y, Cui X, Liao G, Ke C, Xu P, Li X, Zhang C, Yao X, Xu Y, Li T, Su B, Chen Z, Ma R, Jiang Y, Ma X, Bi D, Ma J, Yang H, Li X, Tang L, Yu Y, Wang Y, Song H, Liu H, Wu M, Yang Y, Xue Z, Li L, Li Q, Pang Y. Nontuberculous mycobacterial pulmonary disease and associated risk factors in China: A prospective surveillance study. J Infect. 2021 Jul;83(1):46-53. doi: 10.1016/j.jinf.2021.05.019. Epub 2021 May 25. PMID 34048821
- [Background] Kwak N, Park J, Kim E, Lee CH, Han SK, Yim JJ. Treatment Outcomes of Mycobacterium avium Complex Lung Disease: A Systematic Review and Meta-analysis. Clin Infect Dis. 2017 Oct 1;65(7):1077-1084. doi: 10.1093/cid/cix517. PMID 28582488
- [Background] Diel R, Nienhaus A, Ringshausen FC, Richter E, Welte T, Rabe KF, Loddenkemper R. Microbiologic Outcome of Interventions Against Mycobacterium avium Complex Pulmonary Disease: A Systematic Review. Chest. 2018 Apr;153(4):888-921. doi: 10.1016/j.chest.2018.01.024. Epub 2018 Feb 2. PMID 29410162
- [Background] Magis-Escurra C, Alffenaar JW, Hoefnagels I, Dekhuijzen PN, Boeree MJ, van Ingen J, Aarnoutse RE. Pharmacokinetic studies in patients with nontuberculous mycobacterial lung infections. Int J Antimicrob Agents. 2013 Sep;42(3):256-61. doi: 10.1016/j.ijantimicag.2013.05.007. Epub 2013 Jul 7. PMID 23837923
- [Background] van Ingen J, Aksamit T, Andrejak C, Bottger EC, Cambau E, Daley CL, Griffith DE, Guglielmetti L, Holland SM, Huitt GA, Koh WJ, Lange C, Leitman P, Marras TK, Morimoto K, Olivier KN, Santin M, Stout JE, Thomson R, Tortoli E, Wallace RJ Jr, Winthrop KL, Wagner D; for NTM-NET. Treatment outcome definitions in nontuberculous mycobacterial pulmonary disease: an NTM-NET consensus statement. Eur Respir J. 2018 Mar 22;51(3):1800170. doi: 10.1183/13993003.00170-2018. Print 2018 Mar. No abstract available. PMID 29567726
- [Background] Daley CL, Iaccarino JM, Lange C, Cambau E, Wallace RJ Jr, Andrejak C, Bottger EC, Brozek J, Griffith DE, Guglielmetti L, Huitt GA, Knight SL, Leitman P, Marras TK, Olivier KN, Santin M, Stout JE, Tortoli E, van Ingen J, Wagner D, Winthrop KL. Treatment of nontuberculous mycobacterial pulmonary disease: an official ATS/ERS/ESCMID/IDSA clinical practice guideline. Eur Respir J. 2020 Jul 7;56(1):2000535. doi: 10.1183/13993003.00535-2020. Print 2020 Jul. PMID 32636299
- [Background] Alffenaar JW, Martson AG, Heysell SK, Cho JG, Patanwala A, Burch G, Kim HY, Sturkenboom MGG, Byrne A, Marriott D, Sandaradura I, Tiberi S, Sintchencko V, Srivastava S, Peloquin CA. Therapeutic Drug Monitoring in Non-Tuberculosis Mycobacteria Infections. Clin Pharmacokinet. 2021 Jun;60(6):711-725. doi: 10.1007/s40262-021-01000-6. Epub 2021 Mar 10. PMID 33751415
- [Derived] Zheng X, Wang L, Davies Forsman L, Zhang Y, Chen Y, Luo X, Liu Y, Bruchfeld J, Hu Y, Alffenaar JC, Sha W, Xu B. Correlation of drug exposure and bacterial susceptibility with treatment response for Mycobacterium avium complex lung disease: protocol for a prospective observational cohort study. BMJ Open. 2023 Oct 3;13(10):e075383. doi: 10.1136/bmjopen-2023-075383. PMID 37788924